CLINICAL TRIAL: NCT01618123
Title: The Impact of Short- and Long-term Endothelial Function Assessment by Peripheral Arterial Tonometry (PAT) on Clinical Outcome in Subjects Admitted to Chest Pain Unit (CPU)
Brief Title: Association of Endothelial Function and Clinical Outcomes in Subjects Admitted to Chest Pain Unit
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-9437-MS-CTIL
Record Dates: First submitted 2012-06-10; First posted 2012-06-13 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Myocardial Infarction; Death; Cerebrovascular Accident; Congestive Heart Failure; Angina Pectoris
Keywords: Endothelial function; Coronary disease; Atherosclerosis; Chest pain
MeSH Terms: conditions — Myocardial Infarction; Death; Stroke; Heart Failure; Angina Pectoris; Coronary Disease; Atherosclerosis; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All CPU subjects: All subjects admitted to the CPU with low to moderate probability for CAD and negative troponin, will undergo the following tests upon arrival following clinical evaluation and their consenting to the study: resting ECG, EndoPAT testing and then after stress nuclear imaging or stress echocardiography. Except for EndoPAT testing, all other tests were conducted according to the routine CPU protocol.

SUMMARY:
It is recognized that endothelial dysfunction is a major factor contributing to the atherogenic process. Abnormal function of the endothelium is detectable prior to obvious intimal lesions in patients with risk factors for atherosclerosis. Endothelial dysfunction is a systemic disorder and a key variable in the pathogenesis of atherosclerosis and its complications. Measurement of peripheral vasodilator response with fingertip peripheral arterial tonometry (PAT) technology (EndoPAT; Itamar Medical, Caesarea, Israel) is emerging as a useful method for assessing vascular function. EndoPAT may be a potential valid test increasing the accuracy, sensitivity and specificity for detection of subjects to chest pain unit (CPU) with chest pain but no obvious coronary artery disease (CAD). This is a relatively fast non-invasive bedside test, relatively low-cost and has no side effects. Therefore, the primary objective of the study is to test the hypothesis that abnormal endothelial function as assessed by EndoPAT testing will increase the prediction of the short (in-hospital) and long-term (1-year) outcome of patients presenting to the chest pain unit.

DETAILED DESCRIPTION:
All subjects admitted to the CPU with low to moderate probability for CAD and negative troponin, will undergo the following tests upon arrival following clinical evaluation and their consenting to the study: resting ECG, EndoPAT testing and then after stress nuclear imaging or stress echocardiography. Except for EndoPAT testing, all other tests will be conducted according to the routine CPU protocol.

The results of the EndoPAT will be blinded to the treating physician until the end of the study and all patients will be managed according to the current CPU protocol, including 24-h Holter monitoring, repeat resting ECG and exercise tests (nuclear SPECT imaging or stress echocardiography, whichever is available) in addition to repeat clinical and troponin tests evaluations.

All clinical data of the recruited subjects the will be recorded and evaluated after completion of the study.

Long-term clinical follow-up All patients will be followed by telephone contact after 6 and 12 months for combined major adverse cardiovascular end-points (MACE) which include all-cause mortality, non-fatal myocardial infarction, hospitalization for heart failure or angina pectoris, stroke, coronary artery bypass grafting and percutaneous coronary interventions, by physicians who will be blinded to the patients' baseline clinical status and endothelial function (assessed by EndoPAT) results. All MACE will be validated by review of medical records by senior cardiologists blinded to the endothelial function results. In addition, on-line access to this information will facilitate verification and safe documentation of all events. In addition, written medical records will be reviewed by cardiologists in the event of any death, hospitalization and/or angina pectoris.

At the end of the study the cost effectiveness on prediction of short (in-hospital) and long (6 months, and 1 year) of EndoPAT will be assessed and will be compared to the stress tests (nuclear imaging and/or echocardiography).

ELIGIBILITY:
Inclusion Criteria:

* All subjects admitted to the CPU with low to moderate probability for CAD and negative troponin.

Exclusion Criteria:

* Subjects with chest pain and positive troponin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects admitted to the CPU with low to moderate probability for CAD and negative troponin, will undergo the following tests upon arrival following clinical evaluation and their consenting to the study: resting ECG, EndoPAT testing and then after stress nuclear imaging or stress echocardiography. Except for EndoPAT testing, all other tests were conducted according to the routine CPU protocol.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The association of EndoPat and short-term and long-term outcomes | 1 and 2 years
  To test the hypothesis that abnormal endothelial function as assessed by EndoPAT testing will increase the prediction of the short (in-hospital) and long-term (1-year) outcome of patients presenting to the chest pain unit.

SECONDARY OUTCOMES:
The comparison of different imaging modalities on short- and long-term outcomes | 1 and 2 years
  To compare association of EndoPAT, nuclear SPECT imaging and echocardiographic stress testing on short (in-hospital) and long-term (6 months and 1 year) clinical outcome of patients with chest pain who were admitted to chest pain unit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shechter, MD, Principal Investigator — Chaim Sheba Medical Center; Shlomi Matetzky, MD, Principal Investigator — Chaim Sheba Medical Center; Amir Lerman, MD, Principal Investigator — Mayo Clinic; Joerg Herman, MD, Study Director — Mayo Clinic
Locations (2):
- Mayo Clinic Chest Pain Unit, Emergency Department, Rochester, Minnesota, United States
- Chest Pain Unit, Chaim Sheba Emergency Department, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shechter M, Natanzon SS, Lerman A, Cohn H, Prasad M, Goitein O, Goldkorn R, Naroditsky M, Koren-Morag N, Matetzky S. Endothelial function predicts 5-year adverse outcome in patients hospitalized in an emergency department chest pain unit. J Cardiovasc Med (Hagerstown). 2023 Oct 1;24(10):729-736. doi: 10.2459/JCM.0000000000001502. Epub 2023 May 18. PMID 37222628